CLINICAL TRIAL: NCT02996409
Title: The Value of a High-Volume Image-Guided Injection in Chronic Midportion Achilles Tendinopathy: a Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: High-Volume Image-Guided Injection in Chronic Midportion Achilles Tendinopathy
Acronym: HAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Arthritis Association (Industry); The Anna Foundation (Other)
Responsible Party: Principal Investigator, A.C. van der Vlist, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 51623
Record Dates: First submitted 2016-10-20; First posted 2016-12-19 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Tendinopathy; Achilles Tendon Pain; Injection Site Fibrosis
MeSH Terms: conditions — Tendinopathy | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Volume Image-Guided Injection (Experimental): HVIGI: Injection of 50 cc ( 40 cc 0,9% sodium chloride solution + 10 cc 1% lidocain) in combination with a progressive exercise program and gradual return to sports activities.
  Interventions: Drug: HVIGI; Other: Progressive exercise program
- Low-Volume Image-Guided Injection (Placebo Comparator): LVIGI: Injection of 2 cc (1.6 cc 0.9% Sodium chloride solution + 0.4 cc 1% lidocain) in combination with a progressive exercise program and gradual return to sports activities.
  Interventions: Drug: LVIGI; Other: Progressive exercise program

INTERVENTIONS:
Drug: HVIGI — High Volume Image-Guided Injection with a saline/lidocain solution
  Other Names: Saline 0.9% 40 ml; Lidocain 1.0% 10 ml
  Arms: High-Volume Image-Guided Injection
Drug: LVIGI — Placebo control with injection of a saline/lidocain solution (low volume)
  Other Names: Saline 0.9% 1.6 ml; Lidocain 1.0% 0.4 ml
  Arms: Low-Volume Image-Guided Injection
Other: Progressive exercise program — A 12-week during progressive exercise training program consisting of isometric, isotonic and eccentric calf exercises.

SUMMARY:
Overuse injury of the Achilles tendon is a common entity in athletes. Currently, the usual treatment for chronic midportion Achilles tendinopathy is an eccentric exercise program. In most cases this gives satisfactory results, however there is a significant group of patients in which the exercise program is not sufficient. Prior to our study, three United Kingdom based studies have investigated the efficacy of High-Volume Image-Guided Injections (HVIGI's) in chronic midportion Achilles tendinopathy. They all showed promising results. However none of these studies had an adequate control group. This double-blind, placebo-controlled, randomized clinical trial will investigate the value of a High-Volume Image-Guided Injection in chronic midportion Achilles tendinopathy.

DETAILED DESCRIPTION:
Background of the study - Overuse injury of the Achilles tendon is a common entity in athletes. Especially middle aged athletes are at risk. Elite running athletes have a lifetime risk of sustaining an Achilles tendon injury of 52%. At the moment the usual treatment for chronic midportion Achilles tendinopathy is an excentric exercise program. In most cases this gives great results, however there is a significant group of patients in which the exercise program is not sufficient. Three United Kingdom-based case series evaluated the efficacy of High-Volume Image-Guided Injections (HVIGI's) in chronic midportion Achilles tendinopathy. They all showed promising results. However none of these studies used a comparative group. There is consequently a lack of high-quality studies in this field and therefore the investigators cannot recommend this treatment yet for this indication.

Objective of the study - To investigate the efficacy of a high-volume image guided injection (HVIGI) in chronic midportion Achilles tendinopathy.

Hypothesis - The average VISA-A score is higher in the patient group treated with a progressive exercise program in combination with a high volume image guided injection in comparison with the group treated with low volume injection as a control group in combination with a progressive exercise program.

Study design - A double-blind, randomized, placebo-controlled clinical trial. Randomization and stratification (based on activity level using the Ankle Activity Score) will be performed using a computer-generated model. Measurements will be performed at baseline, 2, 6, 12 and 24 weeks post injection. At every time point both the primary and secondary outcome measurements will be collected. The painDETECT and the Pain Coping Inventory questionnaires will be derived at baseline and 24 week post injection.

Study population - In total, 80 patients with clinically diagnosed chronic midportion Achilles tendinopathy will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years.
2. Clinical diagnosis of chronic midportion Achilles tendinopathy: Painful swelling of the Achilles tendon, 2-7 cm proximal to it's calcaneal insertion.
3. Non-response to exercise program for 6 weeks.
4. Painful Achilles tendon for more than 2 months.
5. Neovascularisation is present on Power Doppler Ultrasonography examination

Exclusion Criteria:

1. Clinical suspicion of insertional disorders (pain at the site of the insertion of the Achilles tendon on the calcaneum)
2. Clinical suspicion of an Achilles tendon rupture (Thompson test abnormal and palpable "gap")
3. Clinical suspicion of plantar flexor tenosynovitis (posteromedial pain when the toes are plantar flexed against resistance)
4. Clinical suspicion of n.suralis pathology (sensitive disorder in the area of the sural nerve)
5. Clinical suspicion of peroneal subluxation (visible luxation of the mm. Peronea spot in combination with localized pain)
6. Suspicion of internal disorders: spondylarthropathy, gout, hyperlipidemia, Rheumatoid Arthritis and sarcoidosis.
7. Condition that prevents the patients from executing an active exercise program
8. Recently prescribed drugs (within 2 years) with a putative effect on symptoms and tendon healing (quinolone antibiotics, corticosteroids).
9. Previous Achilles tendon rupture.
10. Patient has received surgical intervention for his injury.
11. Patient does not wish, for whatever reason, to undergo one of the two treatments
12. A medical condition that would affect safety of injection (e.g. peripheral vascular disease, use of anticoagulant medication)
13. Known presence of a pregnancy
14. Condition of the Achilles tendon caused by medications (arising in relation to moment of intake), such as quinolones and statins
15. Inability to give informed consent.
16. Participation in other concomitant treatment programs.
17. Patient has already one side included in this study.
18. Allergy for lidocain.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment - Achilles questionnaire (VISA-A) | Change in VISA-A score at 24 weeks

SECONDARY OUTCOMES:
Pain detect questionnaire (PD-Q) | Change in pain detect score at 24 weeks
The Pain Coping Inventory (PCI) | Change in PCI score at 24 weeks
10 hop test | Change in visual analogue scale score following a 10 hop test at 24 weeks
Flexibility m. gastrocnemius using a goniometer | Change in flexibility of the gastrocnemius muscle at 24 weeks
Flexibility m. soleus using a goniometer | Change in flexibility of the soleus muscle at 24 weeks
Power m. gastrocnemius using a hand-held dynamometer | Change in power of the gastrocnemius muscle at 24 weeks
Power m. soleus using a hand-held dynamometer | Change in power of the soleus muscle at 24 weeks
Degree of neovascularisation (determined with standardized Power Doppler Ultrasonography examination) | Change in degree of neovascularization at 24 weeks
  Ultrasonography examination before and after eccentric/isotonic calf exercises or rest
Return to sports using a standardized weekly questionnaire | Change in return to sport at 24 weeks
Compliance to the exercise program and return to sports activity program using a standardized weekly questionnaire assessing the percentage of exercises that is performed | Change in compliance at 24 weeks
Patient satisfaction with treatment results | Change at 24 weeks
Patient Acceptable Symptom Scale (PASS) | Change at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: R.J. de Vos, PhD, Principal Investigator — Erasmus MC University Medical Center
Locations (1):
- Erasmus MC University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Oosten CCM, van der Vlist AC, van Veldhoven PLJ, van Oosterom RF, Verhaar JAN, de Vos RJ. Do High-Volume Injections Affect the Ultrasonographic Neovascularization in Chronic Achilles Tendinopathy? A Randomized Placebo-Controlled Clinical Trial. Clin J Sport Med. 2022 Sep 1;32(5):451-457. doi: 10.1097/JSM.0000000000000998. Epub 2021 Dec 9. PMID 36083324
- [Derived] Sleeswijk Visser TSO, van der Vlist AC, van Oosterom RF, van Veldhoven P, Verhaar JAN, de Vos RJ. Impact of chronic Achilles tendinopathy on health-related quality of life, work performance, healthcare utilisation and costs. BMJ Open Sport Exerc Med. 2021 Mar 26;7(1):e001023. doi: 10.1136/bmjsem-2020-001023. eCollection 2021. PMID 33868707
- [Derived] van der Vlist AC, van Oosterom RF, van Veldhoven PLJ, Bierma-Zeinstra SMA, Waarsing JH, Verhaar JAN, de Vos RJ. Effectiveness of a high volume injection as treatment for chronic Achilles tendinopathy: randomised controlled trial. BMJ. 2020 Sep 9;370:m3027. doi: 10.1136/bmj.m3027. PMID 33315586

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT02996409/SAP_001.pdf